CLINICAL TRIAL: NCT06940167
Title: Comparison of the Effectiveness of Kinesio Taping and Myofascial Release in Patients With Cervicogenic Headache
Brief Title: Comparison of Kinesio Taping and Myofascial Release in Cervicogenic Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Fatma CAGLAYAN AGIR, Medical Doctor, Physical Medicine and Rehabilitation, Konya Meram State Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025/5545
Record Dates: First submitted 2025-04-09; First posted 2025-04-23 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Cervicogenic Headache
Keywords: Cervicogenic headache; Myofascial Release; Kinesio taping
MeSH Terms: conditions — Post-Traumatic Headache | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Only the outcomes assessor was blinded to group allocation to reduce measurement bias. Participants and care providers were aware of the intervention being applied.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Myofascial Release Group (Experimental): Group 1 (n=30) will receive myofascial release therapy + home exercise program for four weeks, three sessions per week, totaling 12 sessions.
  Interventions: Other: Myofascial Release Group; Other: Home Exercise Program (Control Group)
- Kinesiology Taping Group (Experimental): Group 2 (n=30) will receive Kinesio taping + home exercise program for four weeks, three sessions per week, totaling 12 sessions
  Interventions: Other: Kinesiology Taping Group; Other: Home Exercise Program (Control Group)
- Home Exercise Group (Experimental): Group 3 (n=30) will receive only a home exercise program for four weeks, three sessions per week, totaling 12 sessions
  Interventions: Other: Home Exercise Program (Control Group)

INTERVENTIONS:
Other: Myofascial Release Group — myofascial release therapy combined with a home exercise program: Myofascial release techniques will be applied manually to the cervical and upper trapezius regions by a trained physiotherapist. The intervention will be administered three times per week for four weeks, totaling 12 sessions. In addition, participants will follow a standardized home exercise program designed to improve cervical mobility and reduce muscle tension.
  Arms: Myofascial Release Group
Other: Kinesiology Taping Group — kinesiology taping combined with a home exercise program : Kinesiology tape will be applied to the cervical region following a standardized taping protocol. The taping will be performed by a trained physiotherapist three times per week for four weeks, totaling 12 sessions. The tape will remain on the skin for 3-5 days per application.
  Arms: Kinesiology Taping Group
Other: Home Exercise Program (Control Group) — Home exercise program: The exercise program includes cervical mobility exercises, stretching, and strengthening exercises aimed at improving posture and reducing muscle tension. The intervention will be performed three times per week for four weeks, totaling 12 sessions.

SUMMARY:
Cervicogenic headache (CGH) is defined as a headache accompanied by neck pain, caused by a disorder in the cervical spine, bones, discs, or soft tissue elements. This study is designed as a prospective, case-control, hospital-based study. A total of 90 patients aged 18-65 years who have been suffering from CGH for at least three months and who present to the Physical Medicine and Rehabilitation Clinic of Meram State Hospital between January 2025 and January 2027 will be included in the study. Patients will be informed about the procedures, and informed consent will be obtained. The study will be conducted in accordance with the Declaration of Helsinki. A detailed medical history will be taken from all participants, and a comprehensive physical examination will be performed. Sociodemographic and clinical characteristics such as age, gender, height, weight, education level, employment status, and income level will be recorded. The 90 CGH patients will be divided into three groups.Group 1 (n=30) will receive myofascial release therapy + home exercise program for four weeks, three sessions per week, totaling 12 sessions. Group 2 (n=30) will receive Kinesio taping + home exercise program for four weeks, three sessions per week, totaling 12 sessions. Group 3 (n=30) will receive only a home exercise program for four weeks, three sessions per week, totaling 12 sessions. All evaluations will be conducted by the same researcher at three time points: before treatment (baseline), at the end of treatment (week 4), and one month after the completion of treatment (week 8).The aim of this prospective clinical study is to compare the effectiveness of Kinesio taping and myofascial release therapy in the treatment of cervicogenic headache.

DETAILED DESCRIPTION:
This randomized, parallel-group clinical trial aims to compare the effectiveness of kinesio taping and myofascial release therapy in patients diagnosed with cervicogenic headache. The study is based on the hypothesis that both interventions can reduce pain intensity and functional disability, but their relative efficacy remains unclear. The trial is designed to provide clinical evidence to guide physiotherapeutic management of cervicogenic headache.

ELIGIBILITY:
Inclusion Criteria:Individuals aged 18-65 years Neck or headache persisting for at least 3 months

Meeting the diagnostic criteria for cervicogenic headache, including:

* Unilateral pain
* Reduced cervical range of motion
* Ipsilateral shoulder discomfort
* Ipsilateral arm discomfort
* Pain exacerbated by different neck movements and tenderness on palpation

Exclusion Criteria:

Migraine Cluster headache Cervical radiculopathy Entrapment neuropathy Myelopathy Rheumatoid arthritis Undergoing cervical spinal surgery Pregnancy Receiving physical therapy within the last 6 months History of major psychiatric disorders History of uncontrolled systemic diseases (cardiovascular, pulmonary, hepatic, renal, hematological, etc.) History of uncontrolled endocrine diseases (e.g., Diabetes Mellitus, hyperthyroidism, etc.)

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Cervicogenic Headache Severity Measured by Visual Analog Scale (VAS) at Baseline, 4 Weeks, and 8 Weeks | Baseline, Week 4 (end of treatment), and Week 8 (1-month follow-up after treatment)
  Headache severity will be assessed using a 10 cm horizontal Visual Analog Scale (VAS), where 0 indicates "no pain" and 10 indicates "worst possible pain." Participants will mark the level of their current headache severity on the scale. Changes will be calculated from baseline to week 4 and week 8.

SECONDARY OUTCOMES:
Change in Headache Impact Test (HIT-6) Score at Baseline, 4 Weeks, and 8 Weeks | Baseline, Week 4, and Week 8
  The HIT-6 is a six-item questionnaire evaluating the impact of headache on daily activities, scored from 36 to 78. Higher scores indicate greater impact.
Change in Headache Disability Index (HDI) Score at Baseline, 4 Weeks, and 8 Weeks | Baseline, Week 4, and Week 8
  The HDI is a 25-item questionnaire assessing the emotional and functional impact of headaches. The total score is used to evaluate disability level.
Change in Quality of Life Measured by Short Form-12 (SF-12) at Baseline, 4 Weeks, and 8 Weeks | Baseline, Week 4, and Week 8
  SF-12 evaluates general health and quality of life across physical and mental domains. Scores are calculated per standard algorithm.
Change in Headache Frequency (Number of Headache Days per Month) at Baseline, 4 Weeks, and 8 Weeks | Baseline, Week 4, and Week 8
  Headache frequency will be recorded using a headache diary. The number of days with headache in the past 4 weeks will be used for assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Meram State Hospital, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) for all primary and secondary outcome measures (e.g., VAS, HIT-6, NDI, SF-12) will be made available to qualified researchers for secondary analysis. Data will be shared upon reasonable request, beginning 6 months after publication, for a period of 3 years. Access will be granted to researchers with methodologically sound proposals by contacting the Principal Investigator via institutional email.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: January 2026 - January 2029
Access Criteria: Qualified researchers with methodologically sound proposals will be able to request access to de-identified individual participant data (IPD), the study protocol, and the statistical analysis plan. Access will be provided upon reasonable request by contacting the Principal Investigator via institutional email. A data sharing agreement may be required before access is granted.